CLINICAL TRIAL: NCT06692946
Title: Evaluation of the Clinical Efficacy of Cooperative Parent-Mediated Therapy (Cooperative-PMT) in Preschool and School-Aged Children With ASD Within the "Autism in Re.Te: Let's Not Leave Them Alone" - Social Project
Brief Title: Clinical Efficacy of Cooperative Parent-Mediated Therapy (C-PMT_in_ASD)
Acronym: C-PMT in ASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ALESSANDRA CARTA (Other)
Collaborators: Bambino Gesù Children's Hospital IRCCS (Other)
Responsible Party: Sponsor-Investigator, ALESSANDRA CARTA, PhD, Università degli Studi di Sassari
Organization: Università degli Studi di Sassari (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Prot. PG/2022/18028; 2021-0545 (Other: Sardinian Foundation)
Record Dates: First submitted 2024-11-06; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Autism Spectrum Disorder; Parent-Training
Keywords: Neurodevelopmental disorders; Parent-child interaction; Community Healthcare service; Additional therapeutic effects
MeSH Terms: conditions — Autism Spectrum Disorder; Neurodevelopmental Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: A rater-blinded RCT conducted in an Italian Child Neuropsychiatry community service. The study included two groups: the experimental CPMT group where children and parents receiving both CPMT and TAU and TAU-CG, where children received only individual PI.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Assessments were not conducted by a blinded independent assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment As Usual (TAU)-Control group (Placebo Comparator): 25 children were randomly assigned to the TAU control group, stratified by cognitive level (IQ or DQ < 70) and language impairment (verbal /non-verbal patients). They undergo Traditional treatement for ASD (CBT and PT).
  Interventions: Behavioral: Treatement as Usual
- Experimental Group: Cooperative parent mediated therapy and Cognitive Behavioural therapy (Experimental): Children were randomly assigned to the experimental group, stratified by cognitive level (IQ or DQ < 70) and language impairment (verbal /non-verbal patients).
  The experimental group consists in 25 children exposed to Cooperative Parent Mediated Therapy as an add on treatment to the TAU (CBT and PT)
  Interventions: Behavioral: Cooperative Parent-Mediated therapy; Behavioral: Treatement as Usual

INTERVENTIONS:
Behavioral: Cooperative Parent-Mediated therapy — Parent-mediated therapy is an intervention where parents are trained to use therapeutic techniques to support their child's development and manage symptoms, often used for conditions like autism spectrum disorder (ASD).
  Other Names: Parent-child training
  Arms: Experimental Group: Cooperative parent mediated therapy and Cognitive Behavioural therapy
Behavioral: Treatement as Usual — Cognitive Behavioral Therapy (CBT) is a structured, short-term psychological treatment that focuses on identifying and changing negative thought patterns and behaviors. It aims to help individuals develop healthier ways of thinking and coping with challenges by addressing both cognitive (thought) and behavioral components.
  Parent training is an educational intervention where parents learn strategies and techniques to effectively manage their child's behavior and support their development, often used to address challenges associated with conditions like autism or ADHD.
  Other Names: Cognitive Behavioral therapy and Traditional Parent Training

SUMMARY:
The research highlights the lack of studies assessing the effectiveness of evidence-based interventions for ASD in community services. This RCT study aims to evaluate the effectiveness of Cooperative Parent Mediated Therapy (CPMT), a parent coaching program previously shown to be effective in tertiary care settings.

DETAILED DESCRIPTION:
Fifty participants with ASD (aged 2-10 years) and their parents were randomized into two groups: both groups received treatment as usual (TAU), but only the experimental group participated in CPMT. The primary outcomes indicated significant improvements in parent-child interaction and benefits in adaptive skills, ASD symptom severity, and parental stress levels in the CPMT group, whereas the TAU group showed no notable changes. The study suggests that the CPMT model is effective in community healthcare settings, representing a significant advancement for ASD therapy.

ELIGIBILITY:
Inclusion Criteria:

* age between 2 and 10 years;
* clinical diagnosis of ASD based on DSM-5 criteria ;
* scores above the autism spectrum cut-off on the Autism Diagnostic Observation Schedule Generic-ADOS-2 ;

Exclusion Criteria:

* 2 years > age < 10 years;
* not received clinical diagnosi for ASD in line with DSM-5 criteria;
* absence of other major medical diagnoses (i.e., epilepsy, genetic syndromes);
* absence of psychosocial treatment during the trial.

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-01-18 (Actual)

PRIMARY OUTCOMES:
parent-child interaction assessed by the PICCOLO scale. | Up to 12months
  parent-child interaction is video recorded and trained observers code-specific parenting behaviors known to predict children's early social, cognitive, and language development.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Alessandra Carta, Sassari
  - Complex Operating Unit of Child and Adolescent Neuropsychiatry - University of Sassari, Sassari

IPD SHARING:
Plan to Share IPD: No
Individual participant data may be shared with other researchers upon specific request and with prior approval from the Ethics Committee.

REFERENCES:
- [Result] Scattoni ML, Fatta LM, Micai M, Sali ME, Bellomo M, Salvitti T, Fulceri F, Castellano A, Molteni M, Gambino G, Posada M, Romano G, Puopolo M. Autism spectrum disorder prevalence in Italy: a nationwide study promoted by the Ministry of Health. Child Adolesc Psychiatry Ment Health. 2023 Oct 28;17(1):125. doi: 10.1186/s13034-023-00673-0. PMID 37898807
- [Result] Autism spectrum disorder in under 19s: support and management. London: National Institute for Health and Care Excellence (NICE); 2021 Jun 14. Available from http://www.ncbi.nlm.nih.gov/books/NBK571989/ PMID 34283415
- [Result] Oono IP, Honey EJ, McConachie H. Parent-mediated early intervention for young children with autism spectrum disorders (ASD). Cochrane Database Syst Rev. 2013 Apr 30;2013(4):CD009774. doi: 10.1002/14651858.CD009774.pub2. PMID 23633377
- [Result] Valeri G, Casula L, Menghini D, Amendola FA, Napoli E, Pasqualetti P, Vicari S. Cooperative parent-mediated therapy for Italian preschool children with autism spectrum disorder: a randomized controlled trial. Eur Child Adolesc Psychiatry. 2020 Jul;29(7):935-946. doi: 10.1007/s00787-019-01395-5. Epub 2019 Sep 23. PMID 31549310